CLINICAL TRIAL: NCT06642441
Title: Effect of Vitamin D Supplementation on Chemotherapy Side Effects After Adjuvant Chemotherapy for Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jiuda Zhao (Other)
Responsible Party: Sponsor-Investigator, Jiuda Zhao, Breast Disease Diagnosis and Treatment Center, Affiliated Hospital of Qinghai University
Organization: Affiliated Hospital of Qinghai University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHQU-2024004
Record Dates: First submitted 2024-10-13; First posted 2024-10-15 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-10

CONDITIONS: Vitamin D; Chemotherapy; Breast Cancer; Adverse Reaction
Keywords: Vitamin D; Breast Cancer; Adverse Reaction
MeSH Terms: conditions — Breast Neoplasms | interventions — Drug Therapy; Ergocalciferols

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chemotherapy + vitamin D2 (Experimental): Before the start of treatment and every 3 weeks thereafter, participants will receive a 10-milligram dose of vitamin D2 injection until adjuvant chemotherapy is completed. They will receive a standard adjuvant chemotherapy regimen, which includes 10 mg of vitamin D2 injections per cycle during treatment. The dosage of adjuvant chemotherapy drugs can be customized according to the clinical judgment of the doctor.
  Interventions: Drug: Chemotherapy + vitamin D2
- chemotherapy (Other): Participants will receive a standard adjuvant chemotherapy regimen for each adjuvant chemotherapy cycle. The dosage of adjuvant chemotherapy drugs can be customized according to the clinical judgment of the doctor.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy + vitamin D2 — Before the start of treatment and every 3 weeks thereafter, participants will receive a 10 mg dose of vitamin D2 injection until adjuvant chemotherapy is completed. They will receive a standard adjuvant chemotherapy regimen, which includes 10 mg of vitamin D2 injections per cycle during treatment. The dosage of adjuvant chemotherapy drugs can be customized according to the clinical judgment of the doctor.
  Arms: Chemotherapy + vitamin D2
Drug: Chemotherapy — Participants will receive a standard adjuvant chemotherapy treatment regimen for each adjuvant chemotherapy cycle. The dosage of adjuvant chemotherapy drugs can be customized according to the clinical judgment of the doctor.
  Arms: chemotherapy

SUMMARY:
This randomized controlled Phase III trial was designed to evaluate the effect of vitamin D supplementation (VD) on chemotherapy side effects following adjuvant chemotherapy in breast cancer

DETAILED DESCRIPTION:
This is a parallel group, open-label randomized controlled trial to investigate the occurrence of side effects of vitamin D supplementation (VD) in adjuvant chemotherapy in patients with breast cancer. Both groups will receive standard adjuvant chemotherapy on day 1 and each subsequent cycle. In addition, vitamin D2 will be given randomly to both groups. Blood samples and imaging results were collected and analyzed before initiation of adjuvant chemotherapy and after every two cycles. The primary outcome to be documented was associated grade III or higher adverse events during adjuvant chemotherapy. Primary and secondary study findings and adverse events will be thoroughly evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years, with an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
2. Primary diagnosis of breast cancer confirmed by preoperative pathological examination.
3. Serum 25(OH)D levels less than 20 ng/ml (50 nmol/L).
4. Patients who have not previously received chemotherapy and who plan to undergo at least 4 cycles of
5. Patients with adjuvant chemotherapy or combined targeted therapy.
6. Life expectancy of at least 6 months.
7. No other uncontrolled benign diseases at the time of recruitment.
8. All patients must have complete clinical medical records.
9. Willingness to voluntarily sign an informed consent form.

Exclusion Criteria:

1. History of invasive breast cancer.
2. Prior systemic treatment for the treatment or prevention of breast cancer.
3. Known allergic reactions to vitamin D or calcium compounds.
4. Comorbidities that may affect vitamin D or calcium balance or bone health.
5. Vitamin D or calcium supplementation in the past 3 months.
6. Presence of other tumors.
7. Pregnant or lactating women.
8. Individuals who do not wish to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and proportion of treatment-related adverse events | 4-6months
  The occurrence of side effects between the two groups from the first to the last chemotherapy

SECONDARY OUTCOMES:
Evaluation of side effects associated with adjuvant therapy (CTCAE v5.0) | From the start of adjuvant therapy to 21 days after the last adjuvant therapy cycle.
  Side effects of adjuvant therapy were evaluated according to CTCAE v5.0 criteria. CTCAE v5.0 was used to evaluate the degree of adverse events after patients received adjuvant chemotherapy. The level of adverse events was divided into 1-5 grades. The higher the level, the more serious the degree of adverse reactions after patients received chemotherapy, and active intervention was required.
Assessment of side effects associated with adjuvant therapy (EQ-5D Health Status Scale) | From the start of adjuvant therapy to 21 days after the last adjuvant therapy cycle.
  Side effects of adjuvant therapy will be assessed according to the EQ-5D Health Status Scale criteria. The EQ-5D health status scale was used to evaluate the health status of patients after chemotherapy. The scale score was between 0 and 1, and the higher the scale score was, the better the health status of patients was reflected
Assessment of side effects associated with adjuvant therapy (Abbreviated Fatigue Scale) | From the start of adjuvant therapy to 21 days after the last adjuvant therapy cycle.
  The side effects of adjuvant therapy will be assessed according to the Concise Fatigue Scale (BFI) criteria, with a score between 0 and 10, with a lower score indicating less fatigue

CONTACTS AND LOCATIONS:
Locations (1):
- Qinghai University Affiliated Hospital, Xining, Qinghai, China